CLINICAL TRIAL: NCT05619900
Title: Registry of Patients Diagnosed With Lysosomal Storage Diseases
Acronym: LSD Registry
Status: Recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 21-34933
Record Dates: First submitted 2022-11-09; First posted 2022-11-17 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Mucopolysaccharidosis I; Mucopolysaccharidosis II; Mucopolysaccharidosis IV A; Mucopolysaccharidosis VI; Mucopolysaccharidosis VII; Pompe Disease Infantile-Onset; Neuronopathic Gaucher Disease; Wolman Disease
Keywords: Lysosomal Storage Disease; LSDs; Inborn Error of Metabolism; Hurler Syndrome; Sly Syndrome; Hunter Syndrome; Mucopolysaccharidosis I; Mucopolysaccharidosis II; Mucopolysaccharidosis IVa; Mucopolysaccharidosis VI; Mucopolysaccharidosis VII; Pompe Disease Infantile-Onset; Neuronopathic Gaucher Disease; Wolman Disease; MPS; Mucopolysaccharidosis
MeSH Terms: conditions — Mucopolysaccharidosis I; Mucopolysaccharidosis II; Mucopolysaccharidosis IV; Mucopolysaccharidosis VI; Mucopolysaccharidosis VII; Gaucher Disease; Wolman Disease; Lysosomal Storage Diseases; Metabolism, Inborn Errors; Mucopolysaccharidoses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Mucopolysaccharidosis I: Prenatally or postnatally diagnosed individuals
  Interventions: Other: There is no intervention
- Mucopolysaccharidosis II: Prenatally or postnatally diagnosed individuals
  Interventions: Other: There is no intervention
- Mucopolysaccharidosis IV A: Prenatally or postnatally diagnosed individuals
  Interventions: Other: There is no intervention
- Mucopolysaccharidosis VI: Prenatally or postnatally diagnosed individuals
  Interventions: Other: There is no intervention
- Mucopolysaccharidosis VII: Prenatally or postnatally diagnosed individuals
  Interventions: Other: There is no intervention
- Infantile-Onset Pompe Disease: Prenatally or postnatally diagnosed individuals
  Interventions: Other: There is no intervention
- Neuronopathic Gaucher: Prenatally or postnatally diagnosed individuals
  Interventions: Other: There is no intervention
- Wolman Disease: Prenatally or postnatally diagnosed individuals
  Interventions: Other: There is no intervention

INTERVENTIONS:
Other: There is no intervention — This is an observational study. There is no intervention. The purpose of the project is to create a database of patients diagnosed either prenatally or after birth with a lysosomal storage disease. The database will be utilized to assess patient outcomes, build on existing clinical management, improve medical decision making, and improve quality of care.

SUMMARY:
This is an international prospective and retrospective registry of patients with Lysosomal Storage Diseases (LSDs) to understand the natural history of the disease and the outcomes of fetal therapies, with the overall goal of improving the prenatal management of patients with LSDs.

DETAILED DESCRIPTION:
The need for methods to track patient outcomes, clinical management, medical decision making, and quality of care are all part of current national mandates in patient safety and quality of care delivery.

The aim of this registry is to prospectively and retrospectively collect data on patients who are diagnosed with Lysosomal Storage Disease and other LSD mutations. Data collected will be used to:

1. Identify patient outcomes of therapies.
2. Improve clinical management of patients with LSDs.
3. Improve medical decision making.
4. Improve quality of care.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 0-64 with a diagnosis of a lysosomal storage disease
* Pregnant patients whose fetus has a diagnosis of a lysosomal storage disease

Exclusion Criteria:

* There are no current exclusion criteria

Max Age: 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Prenatal or postnatal patients diagnosed with a Lysosomal Storage Disease.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-05-31 (Actual); Primary Completion 2050-05-31 (Estimated); Study Completion 2050-05-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with and types of prenatal features of Lysosomal Storage Diseases | 15 years
  Prenatal presentation of symptoms (e.g. hydrops) appearing on fetal imaging such as ultrasound and ECHO.
Number of participants with the presence and levels of glycosaminoglycans (GAGs) in urine. | 15 years
  Laboratory analysis of urine for GAG levels.
Number of participants that show measured levels of antibodies against the enzyme. | 15 years
  Laboratory analysis of blood to measure antibody levels.
Number of participants that show functional cardiac, growth, mobility, and neurocognitive function. | 15 years
  echocardiogram, skeletal survey, neurocognitive assessments such as Bayley III to assess cardiac, growth, mobility and neurocognitive function.

CONTACTS AND LOCATIONS:
Overall Officials: Tippi C MacKenzie, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No